CLINICAL TRIAL: NCT06894667
Title: The Effect of an Antioxidant Gel Compared to Chlorhexidine Gel During the Soft Tissue Healing Process Follow Scaling and Root Planing: A Randomized Controlled Clinical Trial
Brief Title: The Effect of an Antioxidant Gel Compared to Chlorhexidine Gel During the Soft Tissue Healing Process: A Randomized Controlled Clinical Trial
Acronym: Antiox-SRP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, Dr Jagan K Baskaradoss, Associate Professor, Kuwait University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC_816
Record Dates: First submitted 2025-02-23; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Periodontal Diseases
Keywords: Antioxidant; Scaling and root planing
MeSH Terms: conditions — Periodontal Diseases | interventions — Tea Tree Oil

STUDY DESIGN:
Intervention Model Description: A total of 40 subjects would be divided into two groups: Group-1(Control): administration of chlorhexidine gel (n=20) and Group-2 (Test): administration of antioxidant gel (n=20).
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants would be blinded to the intervention and the outcome assessors would also not know the group to which the participant belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): A local gel containing 0.5% chlorhexidene (Curaprox Perioplus Focus Gel,PERIOPLUS+ FORTE, Curaprox, Curaden) would be administered
  Interventions: Drug: Antimicrobial gel
- Test Arm (Experimental): Commercially available antioxidant gel with Tea Tree oil (Tebodont®, Dr. Wild & Co. AG, Basel) would be administered
  Interventions: Drug: Antioxidant gel

INTERVENTIONS:
Drug: Antioxidant gel — An intraoral gel containing Tea Tree oil (Tebodont®, Dr. Wild & Co. AG, Basel) would be applied to the gingival pockets after scaling and root planing
  Other Names: Tea Tree oil (Tebodont®, Dr. Wild & Co. AG, Basel)
  Arms: Test Arm
Drug: Antimicrobial gel — An intraoral gel containing 0.5% Chlorhexidine (PERIOPLUS+ FORTE, Curaprox, Curaden) would be applied to the gingival pockets after scaling and root planing
  Other Names: Chlorhexidine gel (PERIOPLUS+ FORTE, Curaprox, Curaden)
  Arms: Control Arm

SUMMARY:
This study aims to evaluate the comparative impact of chlorhexidine and antioxidant gel on postoperative biomarkers following SRP. By examining biomarkers related to inflammation, oxidative stress, and tissue healing, this research seeks to determine which treatment modality more effectively supports recovery and reduces postoperative complications.

Understanding the differential effects of these interventions on postoperative biomarkers will contribute valuable insights into optimizing SRP outcomes. Correlations between biomarker levels and clinical outcomes, such as periodontal pocket depth and clinical attachment level changes will provide valuable information on the clinical relevance of the findings. This comparison will also guide clinicians in selecting the most appropriate postoperative care to enhance patient recovery and long-term periodontal health.

DETAILED DESCRIPTION:
Background

Periodontitis is characterised by inflammation that results in the loss of periodontal attachment. Scaling and root planing (SRP) is a fundamental non-surgical treatment for periodontitis, which aims to remove the primary causative agents - dental plaque and calculus, from the tooth surfaces. Postoperative care is critical to ensure optimal healing and to manage potential inflammation and microbial load. Traditionally, chlorhexidine, an antimicrobial agent, has been utilized as an adjunctive treatment to prevent infection and manage inflammation following SRP. Chlorhexidine's broad-spectrum antimicrobial properties have been well-documented, and its application has been associated with reduced clinical symptoms and enhanced periodontal healing.

However, recent research has suggested potential benefits of antioxidant gels in promoting tissue repair and reducing oxidative stress, which could be beneficial in the postoperative period. Antioxidant gels, containing compounds such as vitamin C, vitamin E, or polyphenols, are proposed to mitigate oxidative damage and inflammation, potentially offering a different mechanism of action compared to traditional antimicrobial approaches.

Given these advances, there is a need to evaluate and compare the efficacy of chlorhexidine and antioxidant gels in managing postoperative outcomes following SRP. Specifically, assessing their impact on postoperative biomarkers, such as inflammatory cytokines, oxidative stress markers, and periodontal tissue regeneration indicators, could provide valuable insights into their relative effectiveness. In an animal model, found that animals treated with antioxidant gels healed faster and also led to an upregulation of TNFalpha and the antioxidant enzyme superoxide dismutase. However, to the best of our knowledge there are no human clinical studies that have established this relationship. Therefore, this study aims to compare the efficacy adjunctive treatment with chlorhexidine and antioxidant gels along with SRP in the management of patients with periodontitis.

Objectives The objectives of this study are to evaluate and compare the effects of chlorhexidine and antioxidant gel on inflammatory biomarkers (e.g.: Tumor Necrosis Factor-alpha (TNF-alpha); and antioxidant related markers (e.g.: Myeloperoxidase (MPO), among patients undergoing scaling and root planing (SRP). Additionally, the study aims to determine the clinical efficacy of these postoperative treatments in modulating the tissue response.

Methodology Ethics The present study will be performed following the guidelines of the Declaration of Helsinki as revised in 2013 for experimentation involving human patients. All volunteering individuals will be requested to read and sign a consent form written in simple Arabic and English and the study will be presented in accordance with the consolidation standards of reporting trails (CONSORT) guidelines. All participants will be informed that they can withdraw their participation at any phase of the study without consequence. Ethical approval will be obtained from Ethics Committee of Health Science Center at Kuwait University and Ministry of Health. Permission to recruit subjects for this study from the dental clinics of Jaber Hospital has been obtained from the Head of Clinics. The experimental protocol will be also registered at ClinicalTrial.gov.

Study Area/Setting

This prospective study will be conducted between March 2025 and June 2025 at the Dental Clinics of Jaber Hospital and at Kuwait University Dental Center. A convenient sample was selected from regular patients attending the dental clinics.

Grouping Periodontitis is a chronic multifactorial inflammatory disease associated with dysbiotic plaque biofilms and characterised by the progressive destruction of the tooth-supporting apparatus. The definition of periodontitis will be based on the consensus report of Workgroup-4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. Patients with stage III and stage IV periodontitis will be included in this study. A total of 40 subjects would be divided into the following groups: Group-1: administration of chlorhexidine gel (n=20) and Group-2: administration of antioxidant gel (n=20).

The following parameters will be used for the diagnosis of periodontitis: (a) presence of bleeding on gentle probing; (b)probing depth (PD) >6mm; and (c) marginal bone loss (MBL) of at least 3. Patients will be excluded from the study if they present with gingivitis alone, are currently using oral contraceptives, have systemic conditions such as diabetes or cancer, or are smokers (including those who quit within the past 6 months). Additionally, exclusion criteria include recent antibiotic use within the last 3 months, NSAID or bisphosphonate use within the last 90 days, and any use of chlorhexidine in the past 6 months.

Questionnaire A standardized questionnaire will be used to gather information regarding age ( in years ), gender, medical, smoking, and oral health history, including the presence of systemic diseases ( Diabetes mellitus , hypertension ), smoking status, and any recent use of oral contraceptives, antibiotics, NSAIDs, bisphosphonates, or chlorhexidine. This will ensure accurate characterization of the study population and identification of any potential confounding factors. All participants will be asked about their daily tooth brushing habits and the date of the last dental visit and the procedure was done.

Clinical Procedure and Sample Collection All examiners involved in the clinical assessments, laboratory analysis, and statistical evaluations should ideally be blinded to avoid bias. At the initial baseline stage (T0), all participants will undergo non-surgical periodontal therapy, which entails plaque and calculus removal, the use of an ultrasonic scaler, and root planing with sterile curettes (Hu-Freiddy, Chicago, IL, USA). This procedure is expected to last about 60-90 minutes. After the non-surgical therapy, patients will be advised to follow routine oral hygiene practices. Participants will be divided into two groups: one group will receive chlorhexidine gel and the second group will be treated with an antioxidant gel (Tebodont®, Dr. Wild & Co. AG, Basel). They will then be scheduled for a follow-up appointment 4 weeks later (T1).

Salivary Sample Collection The samples during T0 and T1 will be collected from the deepest pocket of the buccal side of the first or second molars as described in an earlier study.

Analysis of Salivary Biomarkers Samples will be stored at -80°C until ready for analysis. TNF-α and MPO will be analyzed using enzyme-linked immunosorbent assay (ELISA) kits from R&D Systems (Minneapolis, MN, USA).

Clinical and Radiographic Examination For all participants, the Löe & Silness gingival index (GI) and Silness & Löe plaque index (PI), bleeding on probing (BOP), and periodontal pocket depth (PD) will be measured on the mesiobuccal, midbuccal, distobuccal, distolingual/palatal, mid-lingual/palatal, and mesio-lingual/palatal surfaces of all maxillary and mandibular teeth by trained and calibrated examiners.

Statistical Analysis Sample size was determined using a computer software G*-power (version 3.0.10; Franz Faul Universitat, Kiel, Germany) based on the values from a previous study 6. It was determined that a sample of 18 individuals/group will be required to get an 80% power and detect the difference in the TNF-α levels between the groups. The Kolmogorov Smirnov-test will be used to assess the data normality and appropriate bivariate and multivariable models will be employed to analyze the data. The level of significance will be set to p<0.05. All the analyses will be carried out using SPSS 27.0 (IBM Corp. Released 2017.IBM SPSS Statistics for Windows, Version 27.0. Armonk, NY: IBM Corp.).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage 3 or 4 periodontitis would be invited to participate in this study.
* The following parameters will be used for the diagnosis of periodontitis: (a) presence of bleeding on gentle probing; (b)probing depth (PD) >6mm; and (c) marginal bone loss (MBL) of at least 3.

Exclusion Criteria:

* Patients will be excluded from the study if they present with gingivitis alone, are currently using oral contraceptives, have systemic conditions such as diabetes or cancer, or are smokers (including those who quit within the past 6 months).
* Recent antibiotic use within the last 3 months, NSAID or bisphosphonate use within the last 90 days, and any use of chlorhexidine in the past 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Plaque Index | baseline
  to assess plaque accumulation
Plaque Index | at 1 month post-intervention
  to assess plaque accumulation
Gingival index | baseline
  for evaluating gingival inflammation
Gingival index | at 1 month post-intervention
  for evaluating gingival inflammation
Probing pocket depth (PPD) | baseline
  for measuring disease severity.PPD is measured in millimetres
Probing pocket depth (PPD) | at 1 month post-intervention
  for measuring disease severity. PPD is measured in millimetres
Clinical attachment level | baseline
  o Clinical attachment level (CAL) is calculated by adding or subtracting probing depth (PD) and gingival recession (GR). The formula is CAL = PD + GR. CAL is measured in millimeters.
Clinical attachment level | at 1 month post-intervention
  Clinical attachment level (CAL) is calculated by adding or subtracting probing depth (PD) and gingival recession (GR). The formula is CAL = PD + GR. CAL is measured in millimeters.
Bleeding on probing (BoP) | baseline
  to assess disease activity
Bleeding on probing (BoP) | at 1 month post-intervention
  to assess disease activity

SECONDARY OUTCOMES:
TNF-α salivary levels | baseline
  TNF-α in micrograms will be analyzed using enzyme-linked immunosorbent assay (ELISA) kits from R&D Systems (Minneapolis, MN, USA).
TNF-α salivary levels | 1 month post intervention
  TNF-α in micrograms will be analyzed using enzyme-linked immunosorbent assay (ELISA) kits from R&D Systems (Minneapolis, MN, USA).
MPO salivary levels | baseline
  MPO in micrograms will be analyzed using enzyme-linked immunosorbent assay (ELISA) kits from R&D Systems (Minneapolis, MN, USA).
MPO salivary levels | 1 month post intervention
  MPO in micrograms will be analyzed using enzyme-linked immunosorbent assay (ELISA) kits from R&D Systems (Minneapolis, MN, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No
The data for the study will be maintained by the Principal investigator.

REFERENCES:
- [Result] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Result] Martin BJ, Campbell PM, Rees TD, Buschang PH. A randomized controlled trial evaluating antioxidant-essential oil gel as a treatment for gingivitis in orthodontic patients. Angle Orthod. 2016 May;86(3):407-12. doi: 10.2319/041515-251.1. Epub 2015 Aug 17. PMID 26280662
- [Result] San Miguel SM, Opperman LA, Allen EP, Svoboda KK. Use of antioxidants in oral healthcare. Compend Contin Educ Dent. 2011 Nov-Dec;32(9):E156-9. PMID 23627309